CLINICAL TRIAL: NCT04355052
Title: An Open-Label Study to Compare the Efficacy, Safety, and Tolerability of Hydroxychloroquine Combined With Azithromycin Compared to Hydroxychloroquine Combined With Camostat Mesylate and to "no Treatment" in Hospitalized Patients Suffering From a Mild or Moderate SARS CoV 2 Virus
Brief Title: Open Label Study to Compare Efficacy, Safety and Tolerability of Hydroxychloroquine Combined With Azithromycin Compared to Hydroxychloroquine Combined With Camostat Mesylate and to "no Treatment" in SARS CoV 2 Virus
Acronym: COSTA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Itsik Levy Dr, Infectious Disease specialist, Sheba Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7092-20-SMC
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: COVID - 19
Keywords: COVID - 19; hydroxychloroquine; camostat mesylate
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; camostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A - HCQ + AZT (Active Comparator): Hydroxychloroquine 400 mg BID on day 1 and than 200 mg BID on days 2-5 + Azithromycin 500 mg QD on day 1 and 250 mg QD on days 2-5
  Interventions: Drug: Hydroxychloroquine in combination of Azithromycin
- B - HCQ + CAM (Experimental): Hydroxychloroquine 400 mg BID on day 1 and than 200 mg BID on days 2-5 + Camostat mesylat 200 mg TID for 10 days
  Interventions: Drug: hydroxychloroquine in combination with camostat mesylate
- C - NI (No Intervention): No Intervention

INTERVENTIONS:
Drug: hydroxychloroquine in combination with camostat mesylate — Two drugs which may act as antivirals against SARS CoVid 2 (Hydroxychloroquine may also act as an immunomodulator, Camostat mesylate is a protease inhibitor)
  Arms: B - HCQ + CAM
Drug: Hydroxychloroquine in combination of Azithromycin — Hydroxychloroquine 400 mg BID on day 1 and than 200 mg BID on days 2-5 + Azithromycin 500 mg QD on day 1 and 250 mg QD on days 2-5
  Arms: A - HCQ + AZT

SUMMARY:
Patients with COVID-19 which are 60 years old or above or with comorbidities are at risk of deteriorating and developing severe illness. This prospective open label study will include people 60 years old or above or younger if at risk for severe disease. Individuals confirmed to have SARS-CoV-2 infection will be identified using medical records screening. They will then be offered to participate in the study and if agree will be given the informed consent. After examining inclusion and exclusion criteria they will be asked to sign the informed consent and after signing Information like immunizations, ECG results, diagnostic images and reports, written medical reports, diagnostic lab testing results (e.g. blood tests, urine tests, blood bank info), allergies and intolerances (drug and food allergies, food intolerances), prescription history, and general patient information (e.g. name, birthdate, personal health number, address, phone number) will be gathered. Those who are not eligible for the study will be informed of the reason(s) for ineligibility (generally it will be a safety exclusion and they should be aware of this). Those who are eligible will be randomized to one of three arms: hydroxychloroquine + azithromycin, hydroxychloroquine + camostat mesylate or "doing nothing" in a ratio of 2:1:2. Study drug will be dispensed by the hospital pharmacy. Follow up will continue for 8 weeks.

DETAILED DESCRIPTION:
This prospective, open-label, placebo-controlled, randomized clinical trial will determine if hydroxychloroquine for 5 days plus camostat mesylate for 10 days, initiated in patients older than 60 years or younger but with risk factors for severe COVID 19 disease will reduce the risk of progression to severe COVID-19 disease compared to hydroxychloroquine plus azithromycin for 5 days or not treating with neither. Severe disease is defined as progression to invasive mechanical ventilation, reduced respiratory parameters (according to NEWS criteria) and 14 and 30-day mortality. This trial will enroll hospitalized consenting adults, who are age 18 or over, have a risk factor for severe disease, have no contraindication to treatment with hydroxychloroquine, can swallow pills, and who do not have severe underlying comorbidity where treatment is not likely to be beneficial to the patient.

The primary outcome will be clinical state of the patient according to NEWS scoring on day 7. Secondary outcomes will be the proportion of participants requiring invasive mechanical ventilation, 14 and 30 -day mortality, and positive viral PCR at day 14.

Randomization will be stratified by age and sex.

Sheba medical center is a tertiary hospital affiliated to Tel Aviv University.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* COVID-19 confirmed by a real-time RT-PCR tests 7 days prior to clinical trial enrollment
* Mild disease (no pneumonia) with at least one of the following risk factors: Age > 55, prior lung or kidney disease, DM with HbA1c > 7.6%, hypertension, CVD, immuno - supressed, organ transplantation, HIV with a CD4 cell count of less than 250 cells/mm3, heavy smoking, BMI > 30.
* Moderate disease - pneumonia, Tachypnea > 24 BPM, tachicardia > 125 BPM, O2 saturation 93% or less

Exclusion Criteria:

* Severe or critical disase
* Assisted ventilation
* Hospitalization in ICU
* Neutrophiles less than 2000
* AST or ALT > 5 times normal
* QTc > 500 msec
* Pregnancy
* Treatment with a drug that prolongs QT

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-04-11 (Actual); Primary Completion 2020-10-11 (Estimated); Study Completion 2020-12-11 (Estimated)

PRIMARY OUTCOMES:
clinical state as reflected by NEWS scoring | 7 days
  the clinical state of the patient regarding respiratory state as defined by the NEWS scoring system
positive PCR | 7 days
  positive PCR SARS COVID 2 in the respiratory system

SECONDARY OUTCOMES:
prevention of ICU | 14 days
  prevention of hospitaliztion in the ICU
prevention of assisted ventilation | 14 days
  prevention of assisted ventilation
prevention of ECMO | 14 days
  prevention of Extracorporeal Membrane Oxygenation (ECMO)
death | 14 days
  death
positive PCR | 14 days
  positive PCR SARS COVID 2 in the respiratory system

OTHER OUTCOMES:
death | 60 days
  death

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Sheba Medical Center, Ramat Gan
  - Sheba Medical Center, Tel Litwinsky